CLINICAL TRIAL: NCT00493480
Title: Danish Carvedilol Study in Portal Hypertension. Carvedilol in the Prevention of Bleeding in Portal Hypertension and Esophageal Varices
Brief Title: Danish Carvedilol Study in Portal Hypertension
Acronym: DACAPO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Erik Feldager/ sponsor, Erik Feldager, Hvidovre Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KF-02-049/03
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Carvedilol; Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carvedilol (Active Comparator)
  Interventions: Drug: carvedilol
- propranolol (Active Comparator): Cirrhotic patients treated with propranolol
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: carvedilol — 6.25 mg of carvedilol for 12 weeks, to achieve a satisfactory pulse reduction the doses are doubled weekly up to a maximum of 25 mg carvedilol daily.
  Arms: carvedilol
Drug: propranolol — 80 mg of propranolol for 12 weeks, to achieve a satisfactory pulse reduction the doses are doubles weekly up to a maximum of 360 mg propranolol daily
  Arms: propranolol

SUMMARY:
Patients with large esophageal varices who have not yet experienced bleeding, are normally treated with propranolol, a beta blocking agent that reduces the portal pressure and thereby diminish the risk of bleeding. 20-40% of the patients do not respond to this treatment or have to discontinue the treatment because of side effects. The aim of this study is to evaluate if carvedilol (a combined alfa -beta blocker) has better efficacy and safety than propranolol in lowering the portal pressure in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* HVPG > 12 mmHg

Exclusion Criteria:

* Respiratory disease that contradict endoscopy
* Hepatic encephalopathy
* Hepatorenal syndrome
* COPD or Asthma
* Treatment with vasoactive drugs within 1 week of inclusion
* Heart disease that contradict treatment with beta-blocking agents
* IDDM
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
If carvedilol is better than propranolol in lowering portal pressure after 3 months of treatment | 3 months

SECONDARY OUTCOMES:
If the effect of a single dose of propranolol can predict the long term effect of propranolol or carvedilol | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Erik F Hansen, MD,Ph.d, Principal Investigator
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Bonefeld K, Hobolth L, Juul A, Moller S. The insulin like growth factor system in cirrhosis. Relation to changes in body composition following adrenoreceptor blockade. Growth Horm IGF Res. 2012 Dec;22(6):212-8. doi: 10.1016/j.ghir.2012.09.001. Epub 2012 Sep 30. PMID 23031335
- [Derived] Hobolth L, Moller S, Gronbaek H, Roelsgaard K, Bendtsen F, Feldager Hansen E. Carvedilol or propranolol in portal hypertension? A randomized comparison. Scand J Gastroenterol. 2012 Apr;47(4):467-74. doi: 10.3109/00365521.2012.666673. Epub 2012 Mar 9. PMID 22401315